CLINICAL TRIAL: NCT01497743
Title: Probiotics in Patients With Moderate-to-severe Distention/ Bloating From Systemic Sclerosis
Acronym: PRISS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KhannaSN0000
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Scleroderma
Keywords: Scleroderma; gastrointestinal; bloating; reflux
MeSH Terms: conditions — Scleroderma, Diffuse; Gastroesophageal Reflux | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Subjects will be randomized into either the probiotic or placebo arm of the study at a 1:1 ratio. All randomized subjects will receive probiotic or matching placebo: 1 capsule orally twice daily, with meals) for the first 4 weeks. There will be a 6-week washout period, followed by 4 weeks of the alternate treatment. The subject will not be on study medication during this washout period.
  Interventions: Drug: Lactobacillus
- Probiotic (Active Comparator): Subjects will be randomized into either the probiotic or placebo arm of the study at a 1:1 ratio. All randomized subjects will receive probiotic or matching placebo: 1 capsule orally twice daily, with meals) for the first 4 weeks. There will be a 6-week washout period, followed by 4 weeks of the alternate treatment. The subject will not be on study medication during this washout period.
  Interventions: Drug: Lactobacillus

INTERVENTIONS:
Drug: Lactobacillus — All randomized subjects will receive probiotic or matching placebo: 1 capsule orally twice daily, with meals) for the first 4 weeks. There will be a 6-week washout period, followed by 4 weeks of the alternate treatment. The subject will not be on study medication during this washout period.
  Other Names: Culturelle

SUMMARY:
Organs of the gastrointestinal tract include the mouth, throat, stomach, intestines, and anus. Patients with scleroderma often have GIT disorders. GIT disorders can be severely debilitating and even life-threatening. Some problems associated with GIT disorders may include heartburn, loss of voice or hoarseness, ulcers (open sores), difficulty swallowing, constipation, diarrhea, malabsorption (impaired absorption of nutrients from the GI tract), diminished peristalsis (decreased in the wavelike motion in the muscles of the intestines), and the inability to control your bowel movements.

Probiotics are the "good bacteria" normally found in your digestive tract. Our group is looking at whether or not taking daily probiotics (lactobacillus) can help alleviate some of these symptoms in scleroderma patients that have GIT disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ≥18 years.
2. Patients with SSc with moderate-to-severe distention/bloating on GIT 2. scale (scale score >1.00).
3. Stable immunosuppressive therapy(ies) for ≥ 1 month.
4. Stable PPI and/or other anti-reflux medications for ≥ 1 month.
5. Stable calcium channel blocker for ≥ 1 month.
6. Stable NSAID for ≥ 1 month.
7. Stable dose of pro-motility agent for ≥ 1 month.

Exclusion criteria:

1. Recent diagnosis for small intestinal bacterial overgrowth (SIBO) during last 1 month.
2. Treatment with antibiotics within last 2 weeks.
3. Currently receiving chemotherapy (pulse cyclophosphamide). It is acceptable to be on methotrexate, mycophenolate mofetil, hydroxychloroquine, or azathioprine.
4. Severe diarrhea (Diarrhea scale score of ≥ 1.01; may suggest untreated SIBO).
5. History of inherited or acquired immunodeficiency

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
1. Proportion of patients with improvement in distention/bloating scale ≥ 0.14 at the end of 4 weeks. A change of 0.14 is the minimally important difference for this scale(9) | 12 months